CLINICAL TRIAL: NCT04950634
Title: Sexual Dimorphism in the Prevalence and Progression of Cardiovascular Autonomic Neuropathy in Patients With Type 1 Diabetes
Brief Title: Sexual Dimorphism in Cardiovascular Autonomic Neuropathy in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: 189/17
Record Dates: First submitted 2021-05-30; First posted 2021-07-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: type1diabetes
Keywords: cardioautonomic neuropathy; sexual dimorphism; subclinical atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Sex might interact with cardioautonomic neuropathy (CAN) in the development of macrovascular disease in patients with type 1 diabetes (T1D). The regulation of the autonomic system shows sexual dimorphism, and may contribute to the cardiovascular risk overload in women with T1D.

The aims of this project are:

A.1) Determining the prevalence of CAN and subclinical atherosclerosis in a large cohort of consecutive patients with T1D as a function of sex (cross-sectional study).

A.2.) Addressing the progression of CAN and subclinical atherosclerosis in patients with T1D as a function of sex (longitudinal prospective study).

A.3.) Investigating the influence of sex steroids and circulating biomarkers in the development and progression of CAN and subclinical atherosclerosis.

Research designs:

A cross-sectional design/prevalence screening study determining the prevalence of CAN as a function of sex in 320 consecutive individuals with DM1.

A longitudinal prospective study: the cohort of prevalence screening study will be prospectively followed, and the assessment of cardiovascular autonomic function and subclinical atherosclerosis will be repeated over time.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of type 1 diabetes mellitus, as defined by ADA criteria

Exclusion Criteria:

* Renal transplantation or renal replacement therapy;
* prior diagnosis of macrovascular disease (CHD, cerebrovascular disease, carotid disease, PAD, or atherosclerotic aortic aneurism);
* ongoing pregnancy;
* diagnosis of types of diabetes mellitus other than type 1;
* diagnosis of types of neuropathy other than diabetic neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are selected from a consecutive cohort of individuals with T1D, who are regularly attending the outpatient clinic of the Diabetes Unit from Hospital Universitario Ramón y Cajal of Madrid.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
To address sexual dimorphism in the prevalence of CAN in patients with T1D. | Two years
  Blood pressure (mmHg) to active standing and Ewing and Clarke tests.
To address sexual dimorphism in the prevalence of CAN in patients with T1D. | Two years
  Heart rate responses (bpm) to active standing and Ewing and Clarke tests.
To address sexual dimorphism in subclinical atherosclerosis in patients with T1D. | Two years
  Mean carotid intima-media thickness (mm)
To assess the role of sex on the progression of cardiovascular dysautonomy in patients with T1D. | Four years
  Blood pressure (mmHg) to active standing and Ewing and Clarke tests.
To assess the role of sex on the progression of cardiovascular dysautonomy in patients with T1D. | Four years
  Heart rate responses (bpm) to active standing and Ewing and Clarke tests.
To assess the role of sex on the progression of subclinical atherosclerosis in patients with T1D. | Four years
  Mean carotid intima-media thickness (mm)

SECONDARY OUTCOMES:
To identify the influence of sex steroids on the evolution of cardiac autonomic dysfunction. | Four years
  Heart rate responses (bpm) to active standing and Ewing and Clarke tests.
To identify the influence of sex steroids on the evolution of cardiac autonomic dysfunction. | Four years
  Blood pressure (mmHg) to active standing and Ewing and Clarke tests.
To identify the influence of sex steroids on the evolution of subclinical atherosclerosis | Four years
  Mean carotid intima-media thickness (mm)
To identify novel circulating markers of CAN | Four years
  Heart rate responses (bpm) to active standing and Ewing and Clarke tests.
To identify novel circulating markers of CAN | Four years
  Blood pressure (mmHg) to active standing and Ewing and Clarke tests.
To identify novel circulating markers of subclinical atherosclerosis | Four years
  Mean carotid intima-media thickness (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Lía Nattero Chávez, Madrid, Madrid, Spain

REFERENCES:
- [Background] Nattero-Chavez L, Insenser M, Amigo N, Samino S, Martinez-Micaelo N, Dorado Avendano B, Quintero Tobar A, Escobar-Morreale HF, Luque-Ramirez M. Quantification of lipoproteins by proton nuclear magnetic resonance spectroscopy (1H-NMRS) improves the prediction of cardiac autonomic dysfunction in patients with type 1 diabetes. J Endocrinol Invest. 2024 Aug;47(8):2075-2085. doi: 10.1007/s40618-023-02289-9. Epub 2024 Jan 6. PMID 38182920
- [Background] Insenser MR, Nattero-Chavez L, Luque-Ramirez M, Quinones SL, Quintero-Tobar A, Samino S, Amigo N, Dorado Avendano B, Fiers T, Escobar-Morreale HF. Investigating the Link between Intermediate Metabolism, Sexual Dimorphism, and Cardiac Autonomic Dysfunction in Patients with Type 1 Diabetes. Metabolites. 2024 Aug 6;14(8):436. doi: 10.3390/metabo14080436. PMID 39195532
- [Background] Nattero-Chavez L, Insenser M, Quintero Tobar A, Fernandez-Duran E, Dorado Avendano B, Fiers T, Kaufman JM, Luque-Ramirez M, Escobar-Morreale HF. Sex differences and sex steroids influence on the presentation and severity of cardiovascular autonomic neuropathy of patients with type 1 diabetes. Cardiovasc Diabetol. 2023 Feb 15;22(1):32. doi: 10.1186/s12933-023-01766-y. PMID 36793089
- [Background] Nattero-Chavez L, Alonso Diaz S, Jimenez-Mendiguchia L, Garcia-Cano A, Fernandez-Duran E, Dorado Avendano B, Escobar-Morreale HF, Luque-Ramirez M. Sexual Dimorphism and Sex Steroids Influence Cardiovascular Autonomic Neuropathy in Patients With Type 1 Diabetes. Diabetes Care. 2019 Nov;42(11):e175-e178. doi: 10.2337/dc19-1375. Epub 2019 Sep 17. No abstract available. PMID 31530659
- See also: Related Info — https://rdcu.be/c5I1C